CLINICAL TRIAL: NCT02814721
Title: Coronal Mode Ultrasound Guided Hemodialysis Cannulation: A Pilot Randomized Comparison With Standard Cannulation Technique
Brief Title: Coronal Mode Ultrasound Guided Hemodialysis Cannulation: Comparison With Standard Cannulation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Analogic Corporation (Industry)
Responsible Party: Principal Investigator, Lalathaksha Kumbar, Senior staff Physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9462
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Arteriovenous Fistula, Cannulation
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard cannulation (No Intervention): The standard cannulation protocol of the center was defined as using 17 gauge needles for the first 3 dialysis sessions, followed by 16 gauge for the next 3, and finally 15 gauge for subsequent sessions.
- Ultrasound guided cannulation (Active Comparator): The study protocol involved similar up titration of needle size over a 3-week period, except that a pre-cannulation evaluation of the fistula was performed using the Sonic Window ultrasound device. The device was used to evaluate and identify the optimal site of cannulation (image 1). Depending upon the cannulator's preference, real-time guidance could be employed during cannulation (image 2, 3). The cannulations were performed by 4 selected personnel trained in device use and successfully completed a competency evaluation on simulator models and a mature dialysis fistula.
  Interventions: Device: Sonic Window ultrasound device

INTERVENTIONS:
Device: Sonic Window ultrasound device
  Arms: Ultrasound guided cannulation

SUMMARY:
Infiltrations from cannulation difficulties result in significant morbidity including loss of vascular access (VA) loss in hemodialysis (HD). Cannulation is reliant on personnel skill and VA characteristics. Surface marking of VA lacks real-time information and traditional ultrasound (US) devices are large, expensive and require skilled operator expertise. Sonic Window© (Analogic Ultrasound, Peabody, MA) is a coronal mode ultrasound device (CMUD) approved for VA cannulation. Study is a single center randomized, prospective pilot study comparing handheld US-guided cannulation of new arteriovenous fistula (AVF) to standard cannulation practices.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease with new arteriovenous fistula being started for cannulation

Exclusion Criteria:

* End-stage renal disease with grafts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GHS West pavilion dialysis center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound Guided Cannulation: The study protocol involved similar up titration of needle size over a 3-week period, except that a pre-cannulation evaluation of the fistula was performed using the Sonic Window ultrasound device. The device was used to evaluate and identify the optimal site of cannulation (image 1). Depending upon the cannulator's preference, real-time guidance could be employed during cannulation (image 2, 3). The cannulations were performed by 4 selected personnel trained in device use and successfully completed a competency evaluation on simulator models and a mature dialysis fistula.
  Sonic Window ultrasound device
Period: Overall Study
Arm/Group | Standard Cannulation | Ultrasound Guided Cannulation
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Cannulation | Ultrasound Guided Cannulation | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.5 [32.5 to 67.5] | 66 [57 to 70] | 61.5 [35.25 to 68.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Infiltration Due to Dialysis Access Cannulation
Description: Infiltration is the extravasation of blood from fistula due to problems with needle insertion into fistula for dialysis.
Time Frame: 3 weeks from use of fistula
Measure: Number; unit: infiltration events
Arm/Group | Standard Cannulation | Ultrasound Guided Cannulation
Number analyzed (Participants) | 4 | 5
infiltration events | 5 | 7

2. Secondary Outcome: Patient Pain Scale
Description: Measured using a scale of 1-10 with 10 being the most severe pain
Time Frame: 3 weeks from use of fistula
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Cannulation | Ultrasound Guided Cannulation
Number analyzed (Participants) | 4 | 5
score on a scale | 2.1 (2.0) | 2.6 (1.8)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Study targeted at a specific intervention of needle insertion only.
Arm/Group | Standard Cannulation | Ultrasound Guided Cannulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No